CLINICAL TRIAL: NCT06663722
Title: A Phase II b Study of Axatilimab in Combination With Extracorporeal Photopheresis (ECP) in Chronic Graft-versus-Host Disease
Brief Title: Axatilimab in Combination With Extracorporeal Photopheresis (ECP) in Chronic Graft-versus-Host Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240116
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Chronic Graft Versus Host Disease; cGVHD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — axatilimab; Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axatilimab in combination with ECP Group (Experimental): Participants in this group will receive Axatilimab in combination with extracorporeal photopheresis (ECP) therapy for up to seven (7) four-week cycles.
  Total participation duration is about 15 months.
  Interventions: Biological: Axatilimab; Procedure: Extracorporeal Photopheresis

INTERVENTIONS:
Biological: Axatilimab — Axatilimab will be administered intravenously (IV) at a dose of 0.3 mg/kg, beginning as a pre-phase dose two weeks prior to initiation of Extracorporeal Photopheresis (ECP) therapy. Thereafter, Axatilimab will be administered with a frequency of one treatment session bi-weekly during each treatment cycle.
Procedure: Extracorporeal Photopheresis — Mandatory ECP therapy will be administered at a frequency of two treatment sessions per week during Cycles 1 through 3, two treatment bi-weekly during Cycles 4 through 6, and two treatments during week 1 of Cycle 7.
  Optional ECP therapy will be administered at a frequency of two treatment sessions during weeks 2 and 4 of Cycles 4 through 6, when mandatory ECP is not administered. Optional ECP therapy will also be administered as two treatment sessions during week 3 of Cycle 7.
  After Cycle 7, participants may receive ECP therapy only at the Investigator's discretion for a maximum Treatment Period of 12 months.
  Other Names: ECP

SUMMARY:
The purpose of this study is to see whether giving participants a combination treatment of Axatilimab and Extracorporeal Photopheresis (ECP) is effective against chronic Graft-versus-Host Disease (cGVHD).

ELIGIBILITY:
Inclusion Criteria:

1. Recipient of allogeneic hematopoietic cell transplantation (HCT).
2. Age greater or equal to 12.
3. Chronic GVHD per 2014 National Institutes of Health Consensus Criteria (NCC) (Jagasia et al. 2015) or overlap syndrome requiring new therapy in patients with at least 2 prior lines of therapy, steroid refractoriness, or steroid dependence:

   1. Prior systemic lines of therapy may include corticosteroids, calcineurin inhibitor (CNI) or sirolimus, or other systemic immunosuppressive agent such as ruxolitinib, belumosudil, or ibrutinib. GVHD prophylaxis does not count as a prior line of therapy.
   2. Steroid refractory is defined as any of the following criteria:

      * i. Manifestations progress despite the use of ≥ 1 mg/kg/day prednisone for at least 1 week
      * ii. Manifestations persist without improvement despite treatment with ≥ 0.5 mg/kg/day or 1 mg/kg every other day for at least four weeks.
      * iii. Recurrence after a CR, or
      * iv. Progression after a PR.
   3. Steroid dependence is defined as inability to control cGVHD symptoms while tapering prednisone below 0.25 mg/kg/day on at least two occasions separated by at least 8 weeks. There must be evidence of clinically active cGVHD.
4. For patients receiving approved or commonly used agents, all GVHD systemic treatments should be discontinued except for corticosteroids and drugs being continued from GVHD prophylaxis at screening.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-3 as assessed at Screening.
6. Platelet count > 50,000 platelets/μL and absolute neutrophil count > 1,000 cells/μL as measured at Screening.
7. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN), unless attributed to presumed cGVHD as measured at Screening.
8. Stable dose of corticosteroids for at least 14 days prior to treatment.
9. Sexually mature individuals must use contraception as described in Section 4.12. For individuals less than 18 years of age, sexual maturity will be determined as per treating pediatrician.

Exclusion Criteria:

1. Pregnancy or breast-feeding.
2. Active relapse of underlying malignancy.
3. History or the presence of interstitial pneumonitis or drug-related pneumonitis.
4. Active gastrointestinal (GI) bleeding.
5. Inability to tolerate volume shifts associated with ECP (e.g., inadequate renal, hepatic, pulmonary and cardiac function (ejection fraction (EF) < 40%) per Investigator discretion.
6. History of myositis.
7. History of splenectomy.
8. History of pancreatitis.
9. History of other malignancy (within 3 years of Screening) unless treated with curative intent and approved by Principal Investigator (PI).
10. Significant, uncontrolled, or active comorbid conditions or are unable to adhere to the study requirements.
11. Acquired Immune Deficiency Syndrome (AIDS) or active hepatitis B (Hep B) or active hepatitis C (Hep C) infection.
12. Prior colony-stimulating factor-1 (CSF-1R) targeted therapies.
13. Prior history of ECP treatment failure or intolerance.
14. Intolerance to methoxsalen, heparin, or citrate products.
15. Patients with aphakia due to risk of increased retinal damage or photosensitive disease (albinism, systemic lupus erythematosus, porphyria).
16. Lack of stable IV access. Acceptable forms include central venous catheter, peripherally inserted central catheter (PICC), or peripheral IV line per institutional guidelines.
17. Insurance denial of coverage for the ECP procedure.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2030-05-05 (Estimated); Study Completion 2030-05-05 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate (ORR) | Up to 24 weeks
  Best overall response rate (ORR) will be reported as the percentage of participants who achieve partial response (PR) or a complete response (CR) to study therapy, as defined by the 2014 National Institutes of Health (NIH) Consensus Development Project on Criteria for Clinical Trials in chronic graft-versus-host disease (cGVHD) while on study treatment.

SECONDARY OUTCOMES:
Proportion of participants experiencing treatment-related adverse events (AEs) | Up to 15 months
  Proportion of participants experiencing treatment-related adverse events (AEs) will be reported. AEs, including serious adverse events (SAEs), will be assessed using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Attribution of AEs and SAEs to study treatment will be reported as possibly, probably and definitely related, as determined by the treating physician.
Proportion of participants experiencing serious adverse events (SAEs) | Up to 15 months
  Proportion of participants experiencing serious adverse events (SAEs) will be reported, regardless of attribution to study treatment, as determined by the treating physician. SAEs will be assessed using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Change in cumulative dose of corticosteroid usage | Baseline, 24 weeks, 1 year
  Change in cumulate dose corticosteroid usage among study participants will be reported, from baseline to 24 weeks and to 1-year post start of Axatilimab. Corticosteroid dosage, recorded as average dose in mg per day, will be recorded at each interval.
Duration of response (DOR) | Up to 15 months
  Duration of response (DOR) is defined as the elapsed time in months from best response (partial response (PR) or complete response (CR)) to documented progression of chronic graft-versus-host disease (cGVHD), start of new therapy, or death for any reason.
Relapse-free survival (RFS) | Up to 15 months
  Relapse-free survival (RFS) is defined as the elapsed time in months from the date of the first dose of study treatment to relapse or recurrence of the primary hematologic malignancy or disorder or death.
Change in Quality of life (QoL) as measured by the modified Lee Symptom Scale (mLSS) score | Baseline, 24 weeks, 1 year
  Changes in quality of life (QoL) from baseline, as measured by the modified Lee Symptom Scale (mLSS) score questionnaire, will be estimated at 24 weeks and 1 year and reported. The mLSS is a 30-item self-reported questionnaire, with seven (7) subscales (skin, eyes, mouth, lung, nutrition, energy and psych) containing 2-7 items which allow calculation of a summary score. Each item uses a 5-point Likert scale ranging from 0 points ("Not at all"/"No symptoms") to 4 points ("Extremely"/"Very severe"). Lower scores indicate improved quality of life. An improvement in > 5-points is considered clinically significant.
Proportion of participants who develop subsequent sclerotic skin disease | Up to 15 months
  The proportion of participants who develop subsequent sclerotic skin disease in those who present without such manifestations will be reported.
Rate of Complete Response (CR) at Best Response | Up to 24 weeks
  The rate of complete response (CR) at best response will be reported as the percentage of patients who achieve CR at best response, as defined by the 2014 National Institutes of Health (NIH) Consensus Development Project on Criteria for Clinical Trials in chronic graft-versus-host disease (cGVHD) while on study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Trent P Wang, DO, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No